CLINICAL TRIAL: NCT04900571
Title: Comparison of Single Antibiotic Paste Nitrofurantoin and Calcium Hydroxide Paste as Intracanal Medicaments in Alleviating Post-Operative Pain in Patients With Symptomatic Irreversible Pulpitis -A Randomized Controlled Trial
Brief Title: Comparison of Nitrofurantoin and Calcium Hydroxide as Intracanal Medicaments in Alleviating Post-operative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nitrofurantoin Vs CaOH
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative; Irreversible Pulpitis
Keywords: Nitrofurantoin; Calcium hydroxide; Intracanal medicaments; Irreversible pulpitis
MeSH Terms: conditions — Pain, Postoperative | interventions — Nitrofurantoin; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nitrofurantoin (Experimental): Measuring pain score using numerical pain scale post-operatively at different time intervals.
  Interventions: Drug: Nitrofurantoin 100 MG
- Calcium Hydroxide (Experimental): Measuring pain score using numerical pain scale post-operatively at different time intervals.
  Interventions: Drug: Nitrofurantoin 100 MG
- Control (Experimental): Measuring pain score using numerical pain scale post-operatively at different time intervals.
  Interventions: Drug: Nitrofurantoin 100 MG

INTERVENTIONS:
Drug: Nitrofurantoin 100 MG — Comparison of alleviating post-operative pain between nitrofurantoin and calcium hydroxide
  Other Names: Calcium Hydroxide

SUMMARY:
Intracanal medicaments have been frequently used in patients with endodontic and periradicular infection for the elimination of microorganisms. Commonly used includes Double Antibiotic Paste, Triple Antibiotic Paste, and Calcium Hydroxide. This study aims to compare the efficacy in alleviating pain between intracanal medicaments Nitrofurantoin and Calcium Hydroxide Paste. 60 patients were randomly divided into 3 groups, each group having 20 patients as following: Group 1: Nitrofurantoin, Group 2: Calcium Hydroxide and Group 3: Control. Preoperative pain was recorded using a numerical pain scale. Pre-operative pain score was initially recorded, followed by Post-operative pain at 12, 24, 48, and 72 hours. Nitrofurantoin has been proven to be an effective intracanal medicament in alleviating immediate post-operative pain in patients with symptomatic irreversible pulpitis as compared to calcium hydroxide.

DETAILED DESCRIPTION:
Intracanal medicaments have been frequently used in patients with endodontic and periradicular infection for the elimination of microorganisms. Commonly used includes Double Antibiotic Paste, Triple Antibiotic Paste, and Calcium Hydroxide. This study aims to compare the efficacy in alleviating pain between intracanal medicaments Nitrofurantoin and Calcium Hydroxide Paste.

60 patients were randomly divided into 3 groups, each group having 20 patients as following: Group 1: Nitrofurantoin, Group 2: Calcium Hydroxide and Group 3: Control. Preoperative pain was recorded using a numerical pain scale. After access preparation, chemomechanical preparation was performed with subsequent placement of intracanal medicaments. Pre-operative pain score was initially recorded, followed by Post-operative pain at 12, 24, 48, and 72 hours, respectively. Root canal treatment was performed in single root teeth with patients suffering from symptomatic irreversible pulpitis.

Total of 20 patients were randomized into 3 groups. Majority of the patients in all 3 groups initially presented with moderate to severe pre-operative pain. After 72 Hours post-operatively, 50% patients in group 1 reported no pain, while 5% patients in both group 2 and 3 had no pain. Pain significantly subsided in group 1 as compared to group 2 and 3. Regarding age and gender, both had no significant relationship with the pain scores in all of the 3 groups.

Nitrofurantoin has been proven to be an effective intracanal medicament in alleviating immediate post-operative pain in patients with symptomatic irreversible pulpitis as compared to calcium hydroxide. While the control group with no intracanal medicament showed little reduction in pain scores. So, nitrofurantoin can be used as a substitute to currently available standard intracanal medicaments.

ELIGIBILITY:
Inclusion Criteria:

* No medical history
* no age restrictions
* no history of allergy to medications used in root canal treatment
* patients suffering from Symptomatic Irreversible Pulpitis

Exclusion Criteria:

* Patients who were not suitable for conventional root canal treatment
* multirooted teeth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Group 1: Nitrofurantoin | 5 months
  Measuring incidence of Post-operative Pain using Numerical Pain Scale
Group 2: Calcium Hydroxide | 5 months
  Measuring incidence of Post-operative Pain using Numerical Pain Scale
Group 3: Control | 5 months
  Measuring incidence of Post-operative Pain using Numerical Pain Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hira Abbasi, BDS, FCPS II Trainee, Principal Investigator — Altamash Institute of Dental Medicine, Pakistan
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan